CLINICAL TRIAL: NCT00462943
Title: A Phase II Open-Label Study of the Subcutaneous Administration of Homoharringtonine. (Omacetaxine Mepesuccinate; OMA) in the Treatment of Patients With Chronic Myeloid. Leukemia (CML) Who Have Failed or Are Intolerant to Tyrosine Kinase Inhibitor Therapy
Brief Title: Open Label Study of Subcutaneous Homoharringtonine (Omacetaxine Mepesuccinate) in Patients With Advanced CML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Cephalon (Industry); ChemGenex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGX-635-CML-203; 2007-001286-15 (EudraCT Number)
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; HHT; Homoharringtonine; Omacetaxine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OMA (Experimental): Omacetaxine mepesuccinate (OMA) Induction: 1.25mg/m^2 subcutaneously twice daily for 14 consecutive days, every 28 days for up to six cycles.
  Omacetaxine mepesuccinate (OMA) Maintenance: 1.25mg/m^2 subcutaneously twice daily for 7 consecutive days, every 28 days for up to 24 months.
  Interventions: Drug: Omacetaxine mepesuccinate

INTERVENTIONS:
Drug: Omacetaxine mepesuccinate — Induction: 1.25mg/m^2 subcutaneously twice daily for 14 consecutive days, every 28 days.
  Maintenance: 1.25mg/m^2 subcutaneously twice daily for 7 consecutive days, every 28 days.
  Response targets during induction vary by chronic myeloid leukemia (CML) subclass (chronic, accelerated, or blast phase). Participants will complete at least one cycle (14 days treatment of a 28 day cycle) of induction therapy before changing to maintenance therapy. Participants not demonstrating evidence of clinical response after 6 induction cycles will be considered for removal from the study.
  Other Names: Homoharringtonine; HHT; Synribo; OMA; CGX-635

SUMMARY:
A Phase II open-label trial of subcutaneous HHT (omacetaxine mepesuccinate) in the treatment of patients who are resistant to or intolerant to Tyrosine Kinase Inhibitors.

DETAILED DESCRIPTION:
This will be an open label, multicenter study of subcutaneous HHT (omacetaxine mepesuccinate) therapy of patients with chronic myeloid leukemia (CML) in chronic, accelerated, or blast phase who have failed or are intolerant to tyrosine kinase inhibitor therapy. Patients will be treated with induction course cycles consisting of subcutaneous (SC) HHT 1.25 mg/m² twice daily for 14 consecutive days every 28 days. Patients will be evaluated every 7 days with complete blood and platelet counts while undergoing induction therapy; the number of consecutive doses of HHT or intervals between subsequent cycles may be adjusted, as clinically indicated, according to guidelines provided in the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 years or older
* Philadelphia chromosome (Ph) positive chronic myelogenous leukemia in either chronic, accelerated, or blast phase
* Patients will have either failed, demonstrated intolerance, or a combination of prior failure and intolerance, to prior treatments with at least two tyrosine kinase inhibitors (TKI's). Failure of TKI treatment may either be primary (never achieved a response) or secondary resistance (loss of response).
* Acceptable Renal and Liver Function
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Sexually active patients and their partners must use an effective double barrier method of contraception

Exclusion Criteria:

* New York Heart Association classification (NYHA) class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition
* Myocardial infarction in the previous 12 weeks.
* Other concurrent illness which would preclude study conduct and assessment
* uncontrolled and active infection, and positive HIV or positive HTLV I/II status, whether on treatment or not.
* Pregnant or lactating.
* Any medical or psychiatric condition, which may compromise the ability to give written informed consent or to comply with the study protocol.
* Lymphoid Ph+ blast crisis
* Patient is enrolled in another clinical investigation within 30 days of enrollment or is receiving another investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03-07 (Actual); Primary Completion 2009-08-04 (Actual); Study Completion 2013-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (29):
- United States (8):
  - Teva Investigational Site 303, Los Angeles, California
  - Teva Investigational Site 308, Beech Grove, Indiana
  - Teva Investigational Site 311, Baltimore, Maryland
  - Teva Investigational Site 305, Buffalo, New York
  - Teva Investigational Site 302, The Bronx, New York
  - Teva Investigational Site 310, Philadelphia, Pennsylvania
  - Teva Investigational Site 301, Houston, Texas
  - Teva Investigational Site 314, Seattle, Washington
- Canada (2):
  - Teva Investigational Site 313, Montreal
  - Teva Investigational Site 309, Toronto
- France (9):
  - Teva Investigational Site 329, Bordeaux
  - Teva Investigational Site 321, Le Chesnay
  - Teva Investigational Site 322, Lille
  - Teva Investigational Site 320, Lyon
  - Teva Investigational Site 324, Nice
  - Teva Investigational Site 328, Paris
  - Teva Investigational Site 323, Poitiers
  - Teva Investigational Site 327, Strasbourg
  - Teva Investigational Site 325, Toulouse
- Germany (2):
  - Teva Investigational Site 331, Berlin
  - Teva Investigational Site 330, Mannheim
- Teva Investigational Site 350, Budapest, Hungary
- India (2):
  - Teva Investigational Site 371, Hyderabad
  - Teva Investigational Site 370, Mumbai
- Teva Investigational Site 390, Bologna, Italy
- Poland (2):
  - Teva Investigational Site 360, Gdansk
  - Teva Investigational Site 361, Warsaw
- Teva Investigational Site 380, Singapore, Singapore
- Teva Investigational Site 340, London, United Kingdom

REFERENCES:
- [Derived] Cortes J, Digumarti R, Parikh PM, Wetzler M, Lipton JH, Hochhaus A, Craig AR, Benichou AC, Nicolini FE, Kantarjian HM; Omacetaxine 203 Study Group. Phase 2 study of subcutaneous omacetaxine mepesuccinate for chronic-phase chronic myeloid leukemia patients resistant to or intolerant of tyrosine kinase inhibitors. Am J Hematol. 2013 May;88(5):350-4. doi: 10.1002/ajh.23408. Epub 2013 Mar 7. PMID 23468307

RESULTS

PARTICIPANT FLOW:
Groups:
- CML: Chronic Phase: Study participants with chronic myeloid leukemia (CML) in the chronic phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
- CML: Accelerated Phase: Study participants with chronic myeloid leukemia (CML) in the accelerated phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
- CML: Blast Phase: Study participants with chronic myeloid leukemia (CML) in the blast phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
Period: Overall Study
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Started | 46 | 31 | 23
Completed | 1 | 1 | 0
Not Completed | 45 | 30 | 23
Not completed — Failure to achieve a response | 5 | 5 | 1
Not completed — Adverse Event | 6 | 4 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Request of Patient, PI, Sponsor or RA | 8 | 2 | 4
Not completed — Disease Progression | 15 | 15 | 9
Not completed — Death | 5 | 2 | 7
Not completed — Stem Cell Transplant | 1 | 1 | 0
Not completed — Bone Marrow Transplant | 1 | 0 | 0
Not completed — Required Lymphocyte Infusion | 1 | 0 | 0
Not completed — Transplant - not specified | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population: all participants who provided written informed consent and received at least 1 dose of study drug constitute the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total
Number analyzed (Participants) | 46 | 31 | 23 | 100
Age, Continuous [Median (Full Range); unit: years] | 58 [20 to 78] | 56 [23 to 71] | 57 [30 to 68] | 57 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 9 | 41
  Male | 26 | 19 | 14 | 59
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31 | 17 | 12 | 60
  Black | 2 | 4 | 5 | 11
  Hispanic | 3 | 2 | 1 | 6
  Asian | 7 | 7 | 4 | 18
  Other | 3 | 1 | 1 | 5
Height [Median (Full Range); unit: centimeter] | 167.7 [155.0 to 188.0] | 167.5 [148.0 to 195.0] | 171.0 [149.9 to 191.0] | 167.6 [148.0 to 195.0]
Weight [Median (Full Range); unit: kilograms] | 79.5 [40.0 to 138.0] | 67.4 [36.5 to 111.8] | 74.0 [41.0 to 136.4] | 74.2 [36.5 to 138.0]
Body Surface Area (BSA) [Median (Full Range); unit: meters^2] | 1.9 [1.3 to 2.5] | 1.7 [1.4 to 2.2] | 1.9 [1.4 to 2.5] | 1.9 [1.3 to 2.5]
New York Heart Association (NYHA) Classification [Number; unit: participants] — * Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  * Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  * Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  * Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bed-bound patients.
  participants
    Class I | 44 | 29 | 23 | 96
    Class II | 2 | 0 | 0 | 2
    Class III | 0 | 0 | 0 | 0
    Class IV | 0 | 0 | 0 | 0
    Not available | 0 | 2 | 0 | 2
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — * Grade 0: Fully active, able to carry on all pre-disease activities without restriction;
  * Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours;
  * Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair.
  participants
    Grade 0 | 27 | 7 | 6 | 40
    Grade 1 | 17 | 19 | 11 | 47
    Grade 2 | 2 | 5 | 5 | 12
    Grade 3 | 0 | 0 | 1 | 1
Time from Initial Chronic Myeloid Leukemia (CML) Diagnosis [Median (Full Range); unit: months] | 74.4 [7.9 to 221.0] | 83.5 [20.3 to 197.1] | 68.7 [6.6 to 195.5] | 74.0 [6.6 to 221.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Overall Hematologic Response by Subpopulation and Total Population
Description: Subpopulations reflect chronic myeloid leukemia (CML) phases at the time of enrollment: chronic, accelerated, and blast phase. Primary endpoints as adjudicated by the Data Monitoring Committee were used for the primary analyses.
  Overall hematologic response for chronic phase participants includes confirmed complete hematologic response (CHR). Overall hematologic response for accelerated or blast phase participants includes confirmed complete hematologic response (CHR), no evidence of leukemia (NEL), or return to chronic phase (RCP). Hematologic response must last >= 8 weeks to be considered meaningful.
  Response rates by disease phase were examined relative to an a priori value of 2.5% using a one-sided lower 95% exact binomial confidence limit. If the lower limit from the one-sided lower 95% confidence limit exceeds 2.5%, the observed response rate will have exceeded the minimum threshold required to demonstrate efficacy.
Time Frame: Day 1 up to 6 months
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total Participants: Treatment included induction therapy of subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
percentage of participants | 67.4 [51.98 to NA] — Lower limit of the 2-sided 95% CI is reported | 25.8 [11.86 to NA] — Lower limit of the 2-sided 95% CI is reported | 8.7 [1.07 to NA] — Lower limit of the 2-sided 95% CI is reported | 41.0 [31.26 to NA] — Lower limit of the 2-sided 95% CI is reported

2. Primary Outcome: Percentage of Participants Achieving a Major Cytogenetic Response by Subpopulation and Total Population
Description: Subpopulations reflect chronic myeloid leukemia (CML) phases at the time of enrollment: chronic, accelerated, and blast phase. Primary endpoints as adjudicated by the Data Monitoring Committee were used for the primary analyses.
  Major cytogenetic response includes complete or partial response. Both confirmed and unconfirmed major cytogenetic response is considered meaningful. Unconfirmed response is based on a single bone marrow cytogenetic evaluation for participants where a confirmatory evaluation is not available.
  Complete response shows 0% Philadelphia chromosome positive (Ph+) cells. A partial response shows >0% - 35% Ph+ cells.
  Response rates by disease phase were examined relative to an a priori value of 2.5% using a one-sided lower 95% exact binomial confidence limit. If the lower limit from the one-sided lower 95% confidence limit exceeds 2.5%, the observed response rate will have exceeded the minimum threshold required to demonstrate efficacy.
Time Frame: Day 1 up to 9 months
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
percentage of participants | 21.7 [10.95 to NA] — Lower limit of the 2-sided 95% CI is reported | 3.2 [0.08 to NA] — Lower limit of the 2-sided 95% CI is reported | 0 [0 to NA] — Lower limit of the 2-sided 95% CI is reported | 11 [5.62 to NA] — Lower limit of the 2-sided 95% CI is reported

3. Secondary Outcome: Percentage of Participants in Each Cytogenetic Response Category Representing the Degree of Suppression of the Philadelphia Chromosome (Ph+)
Description: Cytogenetic response categories:
  * Complete: 0% Ph+ cells
  * Partial: >0%-35% Ph+ cells
  * Minor: >35%-65% Ph+ cells
  * Minimal: >65%-95% Ph+ cells
  * No Response: >95% Ph+ cells
  * Unevaluable: <20 metaphases were examined and/or response could not be assigned
Time Frame: Day 1 up to Month 9
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
percentage of participants
  Complete | 4.3 | 0 | 0 | 2.0
  Partial | 17.4 | 3.2 | 0 | 9.0
  Minor | 8.7 | 9.7 | 0 | 7.0
  Minimal | 6.5 | 6.5 | 4.3 | 6.0
  No Response | 39.1 | 61.3 | 30.4 | 44.0
  Unevaluable | 23.9 | 19.4 | 65.2 | 32.0

4. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Representing the Degree of Suppression of BCR-ABL Transcript Levels Using the Housekeeping Gene GUS
Description: MMR is defined as a ratio of BCR-ABL/standard gene of less than 0.1% according to the international scale. BCR-ABL is a fusion gene of the breakpoint cluster region [BCR] gene and Abelson proto-oncogene [ABL] genes). This analysis used the standard gene GUS. Analysis was performed by quantitative reverse transcription polymerase chain reaction (qRT-PCR) of peripheral blood.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population of participants who had evaluable samples. Participants with no data for these analyses either had degraded samples or the samples were missing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CML: Chronic Phase: Study participants chronic myeloid leukemia (CML) in the chronic phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 22 | 18 | 4 | 44
percentage of participants | 13.6 [2.9 to 34.9] | 0 [NA to NA] — no participants met criteria | 0 [NA to NA] — no participants met criteria | 6.8 [1.4 to 18.7]

5. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Representing the Degree of Suppression of BCR-ABL Transcript Levels Using the Housekeeping Gene ABL
Description: MMR is defined as a ratio of BCR-ABL/standard gene of less than 0.1% according to the international scale. BCR-ABL is a fusion gene of the breakpoint cluster region [BCR] gene and Abelson proto-oncogene [ABL] genes). This analysis used the standard gene ABL. Analysis was performed by quantitative reverse transcription polymerase chain reaction (qRT-PCR) of peripheral blood.
Time Frame: Day 1 up to Month 6
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 38 | 23 | 11 | 72
percentage of participants | 10.5 [2.9 to 24.8] | 4.3 [0.1 to 22.0] | 0 [NA to NA] — no participants met criteria | 6.9 [2.3 to 15.5]

6. Secondary Outcome: Percentage of Participants in Each Hematologic Response Category
Description: Complete Response (CHR)
  * Chronic phase must last at least 8 weeks: WBC <10*10^9/liter, platelets <450*10^9/liter, myelocytes + metamyelocytes <5% in blood, no blasts or promyelocytes in blood, <20% basophils in peripheral blood, no extramedullary involvement.
  * Accelerated and Blast phase must last at least 4 weeks: absolute neutrophil count 1.5*10^9/liter, platelets 100*10^9/liter, no blood blasts, bone marrow blasts <5%, no extramedullary disease.
  Partial Response - CHR plus one or more of the following:
  * Persistence of splenomegaly with a reduction of ≥50% from pre-treatment
  * Platelets > 450*10^9/L
  * Presence of immature cells in the peripheral blood
  * 5% to 25% blasts in the bone marrow
  * If extra-medullary disease pre-treatment, reduction by ≥50% Hematologic Improvement - CHR, except allowing persistent thrombocytopenia (<100*10^9/L), and a few immature cells No evidence of leukemia: Morphologic leukemia-free state, defined as <5% bone marrow blasts.
Time Frame: Day 1 up to Month 6
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
percentage of participants
  Complete response | 67.4 | 19.4 | 8.7 | 39.0
  Partial response | 0 | 3.2 | 0 | 1.0
  Hematologic improvement | 0 | 9.7 | 4.3 | 4.0
  Return to chronic phase | NA — Participants enrolled in chronic phase and therefore cannot respond (improve) to chronic phase. | 6.5 | 0 | 2.0
  No evidence of leukemia | NA — An overall hematologic response for chronic phase participants only included a complete hematologic response. | 0 | 0 | 0
  No response | 21.7 | 58.1 | 78.3 | 46.0
  Unevaluable | 10.9 | 3.2 | 8.7 | 8.0

7. Secondary Outcome: Percentage of Participants With Extramedullary Disease (EMD) at Baseline Achieving a Clinical Response
Description: Clinical response was defined by disease phase and based on evaluations by the independent Data Monitoring Committee (DMC).
  Chronic Phase subgroup: achieving a complete hematologic response and/or major cytogenetic response (complete cytogenetic response or partial cytogenetic response, confirmed or unconfirmed).
  Accelerated Phase and Blast Phase subgroups: achieving complete hematologic response, no evidence of leukemia, return to chronic phase, and/or major cytogenetic response (complete cytogenetic response or partial cytogenetic response, confirmed or unconfirmed).
Time Frame: Day 1 up to Month 9
Population: Intent to treat population of study participants who had extramedullary disease at baseline
Measure: Number; unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 0 | 0 | 2
percentage of participants
  Clinical response |  |  | 0
  Unevaluable |  |  | 50

8. Secondary Outcome: Percentage of Participants With the Largest Percentage Reduction From Baseline of T315I Mutated BCR-ABL
Description: Summarization is based on the best of the individual response assessments. Not assessable indicates that the participant either had no baseline assessment or the % mutation could not be determined in the post-baseline assessment(s).
Time Frame: Day 1 up to Month 9
Population: Intent to treat population of participants with post-baseline assessment of T315I mutated BCR ABL
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 38 | 23 | 11 | 72
percentage of participants
  100% reduction | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  75-99% reduction | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  50-74% reduction | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  25-49% reduction | 0 [0 to 0] | 0 [0 to 0] | 9.1 [0.3 to 52.7] | 1.4 [0.0 to 9.1]
  1-24% reduction | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  0% reduction | 78.9 [76.4 to 100] | 91.3 [83.9 to 100] | 63.3 [47.4 to 99.7] | 80.6 [79.9 to 100]
  Not assessable | 21.1 [NA to NA] — 95% CI not calculated for a non-response category. | 8.7 [NA to NA] — 95% CI not calculated for a non-response category. | 27.3 [NA to NA] — 95% CI not calculated for a non-response category. | 18.1 [NA to NA] — 95% CI not calculated for a non-response category.

9. Secondary Outcome: Number of Treatment Cycles Needed to Achieve Best Hematologic Response
Description: Induction therapy was administered for 14 consecutive days for each 28 days cycle, for up to 6 cycles. All treatment arms were given omacetaxine mepesuccinate via subcutaneous (SC) administration at 1.25 mg/m^2 twice a day (BID) for the 14 consecutive days.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population of participants who had a response to treatment
Measure: Median (Full Range); unit: treatment cycles
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 31 | 8 | 2 | 41
treatment cycles | 1.0 [1 to 5] | 2.0 [1 to 4] | 2.0 [1 to 3] | 1.0 [1 to 5]

10. Secondary Outcome: Number of Treatment Cycles Needed to Achieve Best Cytogenetic Response
Time Frame: Day 1 up to Month 9
Population: Intent to treat population of participants who had a cytogenetic response
Measure: Median (Full Range); unit: treatment cycles
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 17 | 6 | 1 | 24
treatment cycles | 2.0 [1 to 9] | 1.5 [1 to 4] | 1.0 [1 to 1] | 2.0 [1 to 9]

11. Secondary Outcome: Kaplan-Meier Estimates for Time to Onset of Best Hematologic Response
Description: Time to onset was analyzed using Kaplan-Meier estimates. Participants who did not achieve a response are censored at their last visit day.
  Overall hematologic response for chronic phase participants includes confirmed complete hematologic response (CHR). Overall hematologic response for accelerated or blast phase participants includes confirmed complete hematologic response (CHR), no evidence of leukemia (NEL), or return to chronic phase (RCP). Hematologic response must last >= 8 weeks to be considered meaningful.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
months | 1.38 [0.49 to 1.84] | NA [4.14 to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored. | 5.03 [3.13 to NA] — A large percentage of participants were censored.

12. Secondary Outcome: Kaplan-Meier Estimates for Time to Onset of Best Cytogenetic Response
Description: Time to onset was analyzed using Kaplan-Meier estimates. Participants who did not achieve a response are censored at their last visit day.
  Major cytogenetic response includes complete or partial response. Both confirmed and unconfirmed major cytogenetic response is considered meaningful. Unconfirmed response is based on a single bone marrow cytogenetic evaluation for participants where a confirmatory evaluation is not available.
  Complete response shows 0% Philadelphia chromosome positive (Ph+) cells. A partial response shows >0% - 35% Ph+ cells.
Time Frame: Day 1 up to Month 9
Population: Intent to treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 46 | 31 | 23
months | NA [NA to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored.

13. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Subpopulation and Total
Description: TEAE are any untoward events that were newly occurring or worsening from Baseline.
  Treatment related toxicity was considered by the investigator to be unrelated, possibly, probably or unknown related to study drug. Severity was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death. A serious adverse event (SAE) is any untoward medical occurrence that is fatal or life-threatening; results in persistent or significant disability or incapacity; requires or prolongs in-patient hospitalization; is a congenital anomaly/birth defect in the offspring of a patient; and conditions not included in the above that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
  A participant is only counted once in each category (at worst severity or strongest relationship).
Time Frame: up to 4 years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
participants
  >=1 TEAE | 46 | 31 | 23 | 100
  >= 1 SAE | 26 | 19 | 18 | 63
  Worst severity: Grade 1 | 1 | 0 | 0 | 1
  Worst severity: Grade 2 | 4 | 4 | 2 | 10
  Worst severity: Grade 3 | 18 | 6 | 4 | 28
  Worst severity: Grade 4 | 17 | 15 | 6 | 38
  Worst severity: Grade 5 | 6 | 6 | 11 | 23
  Relation to drug: Unrelated | 4 | 4 | 7 | 15
  Relation to drug: Possibly | 5 | 11 | 7 | 23
  Relation to drug: Probably | 36 | 14 | 8 | 58
  Relation to drug: Unknown | 1 | 2 | 1 | 4
  With hematologic toxicity | 36 | 22 | 13 | 71
  Discontinued treatment due to AE | 10 | 11 | 6 | 27
  Deaths during study or follow-up | 35 | 25 | 21 | 71
  Deaths during study (outcome of SAE) | 6 | 6 | 11 | 23

14. Secondary Outcome: Kaplan-Meier Estimates for Duration of Best Hematologic Response
Description: Duration of response is defined as the time from first reported date of hematologic response until the earliest date of objective evidence of disease progression, relapse or death. Data was censored at the last examination date for participants with ongoing response or participants who discontinued treatment for reasons other than adverse event, disease progression or death.
Time Frame: up to four years
Population: Intent to treat population of participants who had a response
Measure: Median (Full Range); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 31 | 8 | 2
months | 7.01 [1.41 to 59.51] | 5.47 [2.40 to 19.70] | 2.67 [1.74 to 3.59]

15. Secondary Outcome: Kaplan-Meier Estimates for Duration of Best Cytogenetic Response
Description: Duration of response is defined as the time from first reported date of cytogenetic response until the earliest date of objective evidence of disease progression, relapse or death. Data was censored at the last examination date for participants with ongoing response or participants who discontinued treatment for reasons other than adverse event, disease progression or death.
Time Frame: up to four years
Population: Intent to treat population of participants who had a response
Measure: Median (Full Range); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 10 | 1 | 0
months | 6.01 [0.92 to 51.94] | 0.07 [0.07 to 0.07] |

16. Secondary Outcome: Kaplan-Meier Estimates for Time to Disease Progression
Description: Time to disease progression is defined as the time from the initiation of treatment until the onset date of death, the development of CML accelerated phase or blast phase, or the loss of complete hematologic response or major cytogenetic response, whichever came first. Participants were censored only if they did not have progression or if they discontinued treatment for reasons other than AE, progression or death.
Time Frame: up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
months | 7.50 [5.86 to 9.64] | 4.84 [3.55 to 6.81] | 2.04 [1.35 to 2.73] | 4.38 [3.55 to 6.45]

17. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival
Description: Overall survival is defined as the time from the initiation of treatment until death from any cause or the last day of participant contact or evaluation for participants that were lost to follow-up. Participants were censored t the last recorded contract or evaluation when a participant was alive at time of analysis. A quarterly phone survey was conducted to collect survival data for participants who discontinued from the study.
Time Frame: up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 46 | 31 | 23 | 100
months | 33.91 [23.75 to NA] — A large percentage of participants were censored | 17.27 [10.56 to 28.45] | 3.52 [2.57 to 5.16] | 17.27 [14.24 to 28.03]

ADVERSE EVENTS:
Time Frame: up to 4 years
Groups:
- Omacetaxine: Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
Arm/Group | Omacetaxine
Serious Adverse Events (participants affected / at risk) | 63/100
Other Adverse Events (participants affected / at risk) | 99/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=100)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 5 (6)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (14)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 8 (8)
Fatigue (General disorders) | 2 (2)
Localised oedema (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (4)
Catheter sepsis (Infections and infestations) | 2 (2)
Injection site infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 3 (4)
Tonsillitis (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=100)
Anaemia (Blood and lymphatic system disorders) | 51 (132)
Bone marrow failure (Blood and lymphatic system disorders) | 6 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 17 (24)
Leukocytosis (Blood and lymphatic system disorders) | 7 (10)
Leukopenia (Blood and lymphatic system disorders) | 13 (55)
Lymphopenia (Blood and lymphatic system disorders) | 8 (20)
Neutropenia (Blood and lymphatic system disorders) | 31 (114)
Thrombocytopenia (Blood and lymphatic system disorders) | 62 (192)
Tachycardia (Cardiac disorders) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (21)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 42 (71)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Gingival bleeding (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 29 (44)
Stomatitis (Gastrointestinal disorders) | 10 (16)
Vomiting (Gastrointestinal disorders) | 17 (22)
Asthenia (General disorders) | 19 (46)
Chills (General disorders) | 10 (13)
Disease progression (General disorders) | 10 (11)
Fatigue (General disorders) | 24 (37)
Injection site erythema (General disorders) | 11 (34)
Injection site rash (General disorders) | 5 (5)
Injection site reaction (General disorders) | 5 (6)
Mucosal inflammation (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 14 (22)
Pyrexia (General disorders) | 28 (50)
Bronchitis (Infections and infestations) | 8 (8)
Cellulitis (Infections and infestations) | 6 (8)
Pneumonia (Infections and infestations) | 13 (15)
Upper respiratory tract infection (Infections and infestations) | 9 (13)
Urinary tract infection (Infections and infestations) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 8 (9)
Alanine aminotransferase increased (Investigations) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 14 (15)
Hyperuricaemia (Metabolism and nutrition disorders) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (18)
Dizziness (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 20 (27)
Insomnia (Psychiatric disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (19)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 7 (8)
Haematoma (Vascular disorders) | 5 (12)
Hypertension (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.